CLINICAL TRIAL: NCT01886950
Title: A Prospective Observational Study to Investigate the Natural History of Bone Histomorphometry and Vascular Calcification in Dialysis-dependent Patients Before and After Renal Transplantation.
Brief Title: Evolution of Bone Histomorphometry and Vascular Calcification Before and After Renal Transplantation
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s52091
Record Dates: First submitted 2013-06-12; First posted 2013-06-26 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Chronic Kidney Disease
Keywords: CKD stage 5; Bone histomorphometry; Renal transplantation
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone biopsy Serum samples A. epigastrica inferior
Oversight: Data Monitoring Committee: No

SUMMARY:
A study of the natural history of bone and mineral disease (BMD) in patients with end-stage renal disease before and after kidney transplantation

DETAILED DESCRIPTION:
Disturbances of mineral and bone diseaeses are frequently observed in CKD patients. Renal osteodystrophy is the term to describe the bone abnormalities. Epidemiological data showed adynamic bone disease (ABD) is the most frequent bone disorder in CKD stage 5D diseases. Low PTH, diabetes mellitus, malnutrition, metabolic acidosis, hypogonadism and low 1,25(OH)2D vitamin D deficiency are known risk factors for ABD. Mounting experimental data point towards a role of protein-bound uremic retention molecules (p-cresyl sulfate and indoxyl sulfate) in the pathogenesis and progression of ABD. ABD is not only recognized as a risk factor for fractures but also for arterial calcification.

The aim of the present study is (1) to investigate the role of indoxyl sulfate and p-cresyl sulfate in the pathogenesis and progression of ABD and arterial calcification in CKD stage5 and (2) to investigate the influence of renal transplantation on bone and arterial metabolism.

ELIGIBILITY:
Inclusion Criteria:

* eligible for renal transplantation and >18 years

Exclusion Criteria:

* use of biphosphonates within the 6 months before the study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: end stage renal disease patients able to consent
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2010-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
bone turnover, as assessed by bone biopsy | at the start of the study
  to investigate the role of indoxyl sulfate and p-cresyl sulfate in the pathogenesis and progression of ABD and arterial calcification in CKD stage5
Evolution of bone turnover, as assessed by bone biopsy | after 1 year
  to evoluation the evolution of bone turnover after succesfull renal transplantation
aortic calcification, as assessed by lumbar X-ray | 1 year
  the assess the evolution of (the degree of) aortic calcification one year after succesfull renal transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Evenepoel, MD,PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven Gasthuisberg, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jorgensen HS, Claes K, Smout D, Naesens M, Kuypers D, D'Haese P, Cavalier E, Evenepoel P. Associations of Changes in Bone Turnover Markers with Change in Bone Mineral Density in Kidney Transplant Patients. Clin J Am Soc Nephrol. 2024 Apr 1;19(4):483-493. doi: 10.2215/CJN.0000000000000368. Epub 2023 Nov 29. PMID 38030558
- [Derived] Jorgensen HS, Behets G, Bammens B, Claes K, Meijers B, Naesens M, Sprangers B, Kuypers DRJ, Cavalier E, D'Haese P, Evenepoel P. Natural History of Bone Disease following Kidney Transplantation. J Am Soc Nephrol. 2022 Mar;33(3):638-652. doi: 10.1681/ASN.2021081081. Epub 2022 Jan 19. PMID 35046132